CLINICAL TRIAL: NCT02529722
Title: Histological and Clinical Biomarkers to Predict the Progression of IgA Nephropathy
Brief Title: Biomarkers for the Progression of IgA Nephropathy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Associate Professor of Medicine, Istanbul University
Other Study IDs: 2907
Record Dates: First submitted 2015-08-07; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: IgA Nephropathy; Glomerular Diseases
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
IgA nephropathy (IgAN) is the most prevalent primary glomerular disease worldwide and an important cause of end stage renal disease. IgAN has an incidence of 8-25 new cases/year/per million age-related population in adults and 3-5/new cases/year/per million age-related population in children and progresses to need of renal replacement treatment in 5-15% at 10 years and in about 20% at 20 years. The variability of the clinical course anticipates different treatment options. There is an absolute need of validated biomarkers to predict risk of progression and indication for treatment at early stages, when lesions can be reversible. This study aimed to evaluate IgAN progression and its histological and clinical correlates.

DETAILED DESCRIPTION:
IgA nephropathy is the most prevalent primary glomerular disease worldwide and an important cause of end stage renal disease. Clinical course varies from long term stable renal functions with minimal proteinuria and microscopic hematuria to rapidly progressive glomerulonephritis with crescents on renal biopsy which progresses to end stage renal disease in a very short time.

In current practice the diagnosis is made with renal biopsy. A less invasive procedure for diagnosis is not present and no serum biomarkers for clinical follow-up, treatment response and prognosis are available. For that reason follow-up of the disease is enabled with indirect markers of renal function like proteinuria, serum creatinine and glomerular filtration rate. These markers are not specific for IgA nephropathy. The lack of disease specific markers hinders the standardization of patient follow-up and treatment. Development of specific and sensitive, repeatable, histopathological and clinical markers for diagnosis, follow up and treatment response in IgA nephropathy the most prevalent primary glomerular disease affecting many patients worldwide will offer prospects of diagnosis and improved prognostication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven IgA nephropathy (defined by standard criteria)
* Patients at all ages will be included regardless of treatment given
* A renal biopsy available for reviewing must include 8 or more glomeruli.
* At least 3 measurements of blood pressure, serum creatinine and proteinuria have to be performed.
* The first measurement should be within 3 months of the date of renal biopsy and the last at the end of the follow-up.
* Patients must comply with the following criteria

  1. have a follow-up longer than 1 year
  2. or having progressed to end-stage renal disease regardless of the duration of follow-up.
* Patients who have received antihypertensive or immunosuppressive medication will be included as well.

Exclusion Criteria:

* Diabetes at the time of first kidney biopsy.
* Solid organ (other than kidney) or bone marrow transplant at the time of biopsy.
* Other pre-existing parenchymal kidney disease on first kidney biopsy, determined by the pathology examination.
* Diagnosis of any of the following diseases from the time of biopsy to the time of enrollment: Systemic lupus erythematosus, HIV infection, active malignancy, except for non-melanoma skin cancer, active hepatitis B or C infection, defined as positive viral load
* Patients with life expectancy < 6 months
* Patients who are unwilling or unable to consent.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the diagnosis of biopsy confirmed IgA nephropathy
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progression to end stage renal disease or two-fold increase in serum creatinine level as compared to baseline | 36 months

SECONDARY OUTCOMES:
Resistance of proteinuria | 36 months
  Resistance of proteinuria defined as no improvement in the daily proteinuria levels or >1 g/24 hr proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University, Istanbul, Turkey (Türkiye)